CLINICAL TRIAL: NCT02031497
Title: Comparison of the Effects of a 12-Week Consumption of Two Carbonated Beverages on Insulin Sensitivity
Acronym: SEDULC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute For European Expertise in Physiology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2012EL0905SEDULC; 120901-10 (Other: ANSM)
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Glucose Homeostasis
Keywords: Sweetener, insulin, body mass index, physical activity
MeSH Terms: conditions — Insulin Resistance; Motor Activity | interventions — Sweetening Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drink with sweeteners (Experimental)
  Interventions: Dietary Supplement: Drink with sweeteners; Dietary Supplement: Drink without sweeteners
- Drink without sweeteners (Active Comparator)
  Interventions: Dietary Supplement: Drink with sweeteners; Dietary Supplement: Drink without sweeteners

INTERVENTIONS:
Dietary Supplement: Drink with sweeteners — Subjects will have to consume a 330ml can of a drink with sweeteners twice per day as part of their usual fluid intake for 12 weeks.
Dietary Supplement: Drink without sweeteners — Subjects will have to consume a 330ml can of a drink without sweeteners twice per day as part of their usual fluid intake for 12 weeks.

SUMMARY:
The purpose of this study is to determine whether consumption of carbonated drinks containing sweeteners affect insulin sensitivity.

DETAILED DESCRIPTION:
Sweeteners are natural or synthetic sugar substitutes which provide a sweetness taste to drink and food with few or no additional calories. Sweeteners are widely used in commercialized beverages. Despite some debate, no significant toxicity was demonstrated at a reasonable level of consumption (less than 20 cans per day). However little data is available on the metabolic effects of a regular consumption of beverages containing sweeteners. The objective of the study is to evaluate the effect of a regular consumption (twice a day for 12 weeks) of a carbonated drink with sweeteners, in a normal diet, compared with unsweetened sparkling water on insulin sensitivity in healthy normoweight and overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Subject taking at least three main meals (breakfast, lunch, dinner)
* Subject able to understand and sign an informed consent
* Subject drinking and enjoying soft drinks
* Subject appreciating sweeteners taste
* 19 kg/m² < BMI< 30 kg/m²

Exclusion Criteria:

* Any severe or acute illness that may influence the results of the study or may be life-threatening
* Pregnant or breastfeeding subject
* Past or present metabolic or digestive diseases, with the exception of a possible appendectomy
* Diabetes or severe acute illness that may alter blood sugar
* Treatment that may interfere with glucose homeostasis
* Past or present kidney disease (renal failure, ... )
* Local or systemic medication that may change water status, metabolism and feeding behavior
* Antiplatelet treatment
* Alcohol consumption ≥ 3-4 glasses / day ( ≥ 21 drinks / week )
* Sustained physical exercise (more than 4 hours per week)
* Subject adding sweeteners (tablets or powder) in their diet
* Subject drinking more than two cans of drinks with sweeteners / day
* Subject dieting to lose weight
* Subject unable or unwilling to consume 2 liters of fluid / day

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Matsuda Insulin sensitivity Index | Before and after each of the two 12-week intervention period

SECONDARY OUTCOMES:
Insulinogenic Index defined as ∆ insulin 0-30 / ∆ glucose 0-30 | Before and after each of the two 12-week intervention period
Disposition index defined as Insulin sensitivity x insulinogenic Index | Before and after each of the two 12-week intervention period
HOMA-IR Index defined as fasting Glycemia x fasting insulinemia/22.5 | Before and after each of the two 12-week intervention period
Dietary intake | Before and after each of the two 12-week intervention period
Physical activity | Before and after each of the two 12-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Bonnet, MD, PhD, Principal Investigator — Centre Hospitalo-Universitaire de Rennes; Fabrice Lainé, MD, PhD, Study Director — Centre Hospitalo-Universitaire de Rennes
Locations (1):
- Unit of Clinical Investigation,Centre Hospitalo-Universitaire de Rennes, Rennes, France

REFERENCES:
- [Derived] Bonnet F, Tavenard A, Esvan M, Laviolle B, Viltard M, Lepicard EM, Laine F. Consumption of a Carbonated Beverage with High-Intensity Sweeteners Has No Effect on Insulin Sensitivity and Secretion in Nondiabetic Adults. J Nutr. 2018 Aug 1;148(8):1293-1299. doi: 10.1093/jn/nxy100. PMID 29982723